CLINICAL TRIAL: NCT03412981
Title: Obesity and Adipose Tissue Inflammation in Pregnant Mothers
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Other Study IDs: 2004215 Pregnant Moms
Record Dates: First submitted 2018-01-20; First posted 2018-01-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pregnant mothers — we will be collecting data on a cohort of pregnant mothers

SUMMARY:
To date very little research has been conducted on pregnant mothers. Research shows that mothers with obesity and gestational diabetes have children who have a higher risk of later developing obesity and diabetes compared to children born to non-obese mothers but the mechanisms are not known. The maternal environment may place these babies at greater risk and it is possible that fat tissue (adipose tissue) releases many chemicals (adipokines and inflammatory cytokines) which may have an impact on the baby. Mothers who have greater amounts of adipose tissue most likely release these adipokines into the baby and it may affect the baby's body composition and/or health.

This project will establish if there is a relationship between obesity and adipose tissue inflammation in pregnant mothers, and if there is a link between inflammation and the child's body composition.

We will recruit mothers with low risk pregnancies already schedule for a C section at about 36 wk. We will do initial testing at 36 wk, adipose tissue collection at delivery, and conduct post testing at 1 month postpartum on the mother and the baby.

DETAILED DESCRIPTION:
Study 1 Visit 1: Sign consent form, age, height, weight, and completion of questionnaires (e.g. food record). Consent will allow the investigators to gain access to medical record to record pregnancy-related health information on the mother (e.g., prenatal care including but not limited to maternal vital signs, clinical documents and fetal well-being - such as # pregnancies; reason for scheduled C-section; starting body weight and weight gain during pregnancy; BP throughout pregnancy; glucose challenge test (GCT) and glucose tolerance test (GTT) results; disease history; medications; pregnancy complications). The investigators will also access any fetal monitoring (e.g., including any cardiac ultrasounds that may have been performed.) Screening fasting bloods - glucose, insulin, HbA1c, blood lipids, CRP, inflammatory cytokine panel (TNFa, IL-6, IL-4, IL-13), adipokines (adiponectin, leptin), and sex hormones (e.g., estradiol, testosterone, progesterone). The investigators will also perform a limited ultrasound to assess fetal cardiac function and adiposity at this time. Subjects will be given a physical activity monitor to wear for 7 days.

Visit 2: C-section: At this visit during the C-section, a sample (~1000 mg/depot) of omental and subcutaneous fat samples will be taken for assessment of inflammatory genes/proteins. Cord blood (~15 ml) for assessment of inflammatory genes/proteins.

Visit 3: 1 month post-partum Mother: Resting blood pressure, fasting blood sample (glucose, insulin, HbA1c, blood lipids, CRP, inflammatory cytokine panel (TNFa, IL-6, IL-4, IL-13), adipokines (adiponectin, leptin)), sex hormones (estradiol, progesterone, testosterone), and body composition measurement. Completion of questionnaires. Subjects will be given a physical activity monitor to wear for 7 days.

Study 2 Women will only be recruited to complete the C-section as described above They will have the option to have the baby measured in the pea pod and to wear a physical activity monitor for a week in the month before delivery.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have low risk pregnancies (21-40 years) and are already scheduled to have a C-section. BMI ≤ 40 kg/m2

Exclusion Criteria:

* We will exclude emergency C-sections
* Subjects will have had a screening ultrasound that demonstrated the absence of congenital anomalies as part of routine prenatal care
* Mothers with high risk pregnancy
* BMI > 40 kg/m2

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on being able to get pregnant
Study Population: Recruiting from women who will deliver their babies at Women and Children's hospital in Columbia, MO
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
TNFa | at delivery
  TNFa, IL-6, IL-4, IL-13

SECONDARY OUTCOMES:
body fat | after delivery
  body composition of the baby
IL-6 | at delivery
  IL-6in abdominal fat
IL-4 | at delivery
  Il-4in abdominal fat
IL-13 | at delivery
  IL-13 in abdominal fat
baby weight | at birth
  kg

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - University of Misouri, Columbia, Missouri
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No